CLINICAL TRIAL: NCT03659357
Title: A Prospective Comparison of Diagnostic Efficacy and Radiomics Study in the Diagnosis and Therapeutic Efficacy Evaluation of Small Bowel Tumor With Dual-phase Enhanced Computed Tomography (CTE) and Magnetic Resonance Enterography (MRE)
Brief Title: Study of Small Bowel Tumor With Dual-phase Enhanced Computed Tomography (CTE) and Magnetic Resonance Enterography (MRE)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJ-IRB20180508
Record Dates: First submitted 2018-08-19; First posted 2018-09-06 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Intestinal Neoplasms
MeSH Terms: conditions — Intestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A-first CTE examination
- B-first MRE examination

SUMMARY:
Purpose: To compare the accuracies of computed tomographic (CT) enterography and magnetic resonance (MR) enterography for the detection and radiomics characterization of small-bowel tumors (including gastrointestinal stromal tumors, adenomas and lymphomas, etc); Hypothesis: MR enterography was noninferior to CT enterography for the diagnosis and evaluation of small bowel tumors in generally well-distended small bowel.

DETAILED DESCRIPTION:
The investigators will conduct a 36-month clinical trial, the specific process is as follows:

1. Incorporate patients with the above criteria, communicate with the participants to make informed consent and sign informed consent;
2. It is recommended that the attending physician issue the corresponding MRE checklist and the CTE checklist and make an appointment to check the same day to remind the patient to perform the corresponding bowel preparation work in advance, and perform renal function tests within 3 days before the examination;
3. The enrolled patients were measured for height and weight, and the BMI was calculated. CTE and MRE were performed according to the results of balanced randomization. The MRE was performed on a 3.0T MRI scanner; the CTE examination was performed on a 320-row CT scanner, and the iodine-containing contrast agent was administered according to the patient's height and weight and GFR;
4. Both examinations require an empty stomach preparation (more than 4 hours), and oral (1500ml) 2.5% mannitol aqueous solution before the examination to ensure intestinal filling, subcutaneous indwelling needle preparation, in order to save patient examination time, so the two examinations are completed within 6 hours, before the second inspection, you need to add 150-300ml of 2.5% mannitol aqueous solution;
5. The images obtained were evaluated by two imaging physicians for lesions, numbers, size changes, density/signal values, and peripheral tissue lesions obtained by the two methods;
6. After the patient has obtained a definitive diagnosis according to the routine medical procedure, the above imaging diagnosis results are compared with the confirmed diagnosis results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical suspicion of small intestinal neoplasms and prescribed CTE and/or MRE examinations;
* Age/sex: unlimited;
* Patients with no severe heart, liver, kidney insufficiency;
* Patients who voluntarily participate in clinical trials and sign written informed consent.

Exclusion Criteria:

* patients with heart and liver insufficiency;
* patients with pacemakers installed and which materials are unknown, and patients with metal implants in the body, and nerve stimulators;
* patients who are allergic to iodine and intestinal contrast agents;
* pregnant women, patients with acute or chronic renal failure and hemodynamic instability;
* patients unable to tolerate adequate breath holding for complete CT or MR examination;
* patients who can not maintain compliance and cannot strictly implement the plan.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients who were suspected of having small bowel tumors on the basis of clinical findings and who were previously diagnosed with small bowel tumors underwent CT and MR enterography.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
the size in centimeters | through study completion, an average of 3 years, the size of the small bowel tumor will be reported.
  the size of the small bowel tumor

SECONDARY OUTCOMES:
volume in cm^3 | through study completion, an average of 3 years
  the volume of the small bowel tumor
intensity of the neoplasms measured in the MRE | through study completion, an average of 3 years
  the intensity of the small bowel tumor measured in the MRE, and it is graded into low, moderate and high.
intensity of the neoplasms measured in the CTE in Hu | through study completion, an average of 3 years
  the intensity of the small bowel tumor measured in the CTE

CONTACTS AND LOCATIONS:
Overall Officials: Yaqi Shen, doctor, Study Chair — Tongji Hospital
Locations (1):
- Yaqi Shen, Wuhan, Hubei, China